CLINICAL TRIAL: NCT01734824
Title: Treatment of Atraumatic Bone Marrow Edema With Denosumab and Teriparatide vs Placebo
Status: Suspended | Phase: Phase 4 | Type: Interventional
Why Stopped: no patients randomized
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Dr. Christian Muschitz, Principal Investigator, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Vinforce-012; Bone marrow edema (Other: Medical Uiversity Vienna - Vinforce)
Record Dates: First submitted 2012-06-02; First posted 2012-11-28 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Bone Marrow Oedema Syndrome; High Turnover Bone Disease; Quality of Life
Keywords: bone marrow edema, denosumab, PTH 1-84
MeSH Terms: interventions — Denosumab; Teriparatide; Parathyroid Hormone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Teriparatide (Active Comparator): daily subcutaneous injection of teriparatide 20µg for three months
  Interventions: Drug: Teriparatide
- Placebo Teriparatide (Placebo Comparator): daily subcutaneous teriparatide placebo injection
  Interventions: Drug: Placebo Teriparatide
- Denosumab (Active Comparator): one subcutaneous injection of denosumab
  Interventions: Drug: Denosumab
- Placebo Denosumab (Active Comparator): one subcutaneous injection of denosumab placebo
  Interventions: Drug: Placebo Denosumab

INTERVENTIONS:
Drug: Denosumab — sc RANKL-inhibitor
  Other Names: Prolia
  Arms: Denosumab
Drug: Teriparatide — daily subcutaneous injection of teriparatide
  Other Names: PTH 1-34
  Arms: Teriparatide
Drug: Placebo Denosumab — one subcutaneous injection denosumab placebo
  Other Names: Prolia
  Arms: Placebo Denosumab
Drug: Placebo Teriparatide — daily subcutaneous placebo injection
  Other Names: PTH 1-34
  Arms: Placebo Teriparatide

SUMMARY:
The etiology of bone marrow edema (BME) is still uncertain. Several studies report therapeutic success with antiresorptive drugs.

This study investigates antiresorptive and osteoanabolic drugs versus placebo in BME

DETAILED DESCRIPTION:
Patients are assigned to receive either denosumab 60mg sc (once) or placebo or daily teriparatide sc for three months or placebo.

MRI examinations at baseline and after three months will be performed. Serum bone turnover markers will be evaluated as well as QoL questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* MRI diagnosed bone marrow edema

Exclusion Criteria:

* any prior antiresorptive or osteoanabolic treatment
* any prior therapy with strontium ranelate
* Hyper-/hypocalcemia
* malignancies
* pregnancy
* and contraindication against denosumab or teriparatide

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2012-05; Primary Completion 2015-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Reduction/termination of bone marrow edema with antiresorptive and osteoanabolic drugs | baseline - month 1 - month 3
  MRI examination, fasting serum levels of bone turnover markers, QoL-questionnaire, VAS score

CONTACTS AND LOCATIONS:
Overall Officials: Christian Muschitz, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University Vienna - St. Vincent Hospital, Vienna, Vienna, Austria